CLINICAL TRIAL: NCT04516382
Title: An Open-label Crossover Study Evaluating the Pharmacokinetics and Pharmacodynamics of Different PTG-300 Regimens in Healthy Volunteers
Brief Title: Pharmacokinetics and Pharmacodynamics of Different PTG-300 Regimens in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Protagonist Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PTG-300-07
Record Dates: First submitted 2020-08-10; First posted 2020-08-18 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: Single group of subjects will sequentially receive PTG-300 as IV, subcutaneous, and intramuscular administration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Intravenous (Experimental): PTG-300 Intravenous
  Interventions: Drug: PTG-300
- Subcutaneous Low Concentration (Experimental): PTG-300 Subcutaneous Low Concentration
  Interventions: Drug: PTG-300
- Subcutaneous High Concentration (Experimental): PTG-300 Subcutaneous High Concentration
  Interventions: Drug: PTG-300
- Intramuscular (Experimental): PTG-300 Intramuscular
  Interventions: Drug: PTG-300

INTERVENTIONS:
Drug: PTG-300 — Active drug

SUMMARY:
To estimate the bioavailability of PTG-300 following subcutaneous and intramuscular administration in healthy volunteers.

DETAILED DESCRIPTION:
This is a single center, open-label study in healthy males. Subjects will be screened for eligibility within 28 days of dosing.

Twelve subjects will receive single doses of the following treatments in a fixed sequence:

Treatment A: Intravenous injection of 1.5 mg PTG-300. Treatment B: 40 mg (40 mg/mL) PTG-300 administered subcutaneously. Treatment C: 40 mg (200 mg/mL) PTG-300 administered subcutaneously. Treatment D: 40 mg (40 mg/mL) PTG-300 administered intramuscularly.

There will be a washout period of at least 7 days between Treatment A and Treatment B and at least 12 days between Treatments B, C, and D.

Subjects' safety will be monitored, and blood samples will be collected for pharmacokinetics and pharmacodynamics (serum iron, serum ferritin, serum transferrin, and transferrin saturation [TSAT]).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers, age 18 to 65 years, inclusive.
2. Subjects must have a Body Mass Index (BMI) between 18 and 32 kg/m2 inclusive.
3. Subjects must have clinical laboratory values within normal range as specified by the testing laboratory, unless deemed not clinically significant by the Investigator.
4. Agree to use a barrier method of contraception from Day -2 to 90 days after the last dose of study drug.
5. Subjects must have the ability and willingness to attend the necessary visits to the study center.

Exclusion Criteria:

1. History of clinically significant endocrine, neurological, gastrointestinal, cardiovascular, haematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases.
2. History of malignancy, with the exception of adequately treated non-melanomatous skin carcinoma.
3. Mentally or legally incapacitated, has significant emotional problems at the time of Screening Visit or expected during the conduct of the study, or has a history of a clinically significant psychiatric disorder that would impact the subjects ability to participate in the trial according to the Investigator.
4. Fever (body temperature >38°C) or symptomatic viral or bacterial infection within 2 weeks prior to screening; evidence of intestinal infection within 30 days prior to screening.
5. History of severe allergic or anaphylactic reactions.
6. A supine blood pressure outside the range of 90 to 139 mm Hg systolic and 50 to 89 mm Hg diastolic, OR heart rate (HR) >100 beats per minute at Screening and at Day -1.
7. Laboratory values that are outside the normal range and considered clinically significant by the Investigator.
8. Positive test for hepatitis C antibody, hepatitis B surface antigen or human immunodeficiency virus (HIV) antibody at Screening.
9. Subjects considered at high risk of iron deficiency according to the Investigator.
10. Subjects with iron deficiency as defined by a ferritin or transferrin saturation below the normal range
11. Clinically significant abnormality on ECG performed at the Screening Visit or prior to administration of the initial dose of study drug.
12. Corrected QT (QTcF) greater than 450 msec at Screening.
13. Subjects with a positive toxicology screening panel.
14. Subjects with a history of substance abuse or dependency or history of recreational IV drug use (by self-declaration).
15. Consumption of >14 alcohol units per week (where 1 unit = 284 mL of beer, 25 mL of 40% spirit, or a 125 mL glass of wine).
16. Unable to refrain from or anticipates the use of any medications, including prescription and non-prescription drugs and herbal remedies (such as St. John's Wort [Hypericum perforatum]), beginning 14 days (or 5 half lives, whichever is longer) before administration of the initial dose of study drug and continuing throughout the study until the final study visit.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — male
Enrollment: 12 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Bioavailability of PTG-300 | Week 1
  Bioavailability (area under the plasma-concentration time) of PTG-300 following subcutaneous and intramuscular administration in healthy volunteers

SECONDARY OUTCOMES:
Serum Iron Pharmacodynamics of PTG-300 | Week 1
  Change from baseline in serum iron following subcutaneous and intramuscular administration in healthy volunteers
TSAT Pharmacodynamics of PTG-300 | Week 1
  Change from baseline in transferrin saturation (TSAT) following subcutaneous and intramuscular administration in healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Protagonist Therapeutics, Inc.
Locations (1):
- Protagonist Clinical Center, Melbourne, Australia